CLINICAL TRIAL: NCT06418763
Title: The Effects of Fermented Brown Seaweed Intake on Glucose Metabolism and Gut Health: a Short-term Study in Healthy Subjects
Brief Title: The Effects of Fermented Brown Seaweed Intake on Glucose Metabolism and Gut Health
Acronym: SEAPRO01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Collaborators: Lund University (Other); Carbiotix AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SEAPRO01
Record Dates: First submitted 2024-04-23; First posted 2024-05-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects
Keywords: seaweed; blood glucose; gut microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baobab spread mixed with fermented seaweed (Active Comparator): Daily intake 2x 15g The product is available as a spread and will be consumed with bread
  Interventions: Dietary Supplement: Baobab spread mixed with fermented brown seaweed
- Baobab spread (Placebo Comparator): Daily intake 2x 15g The product is available as a spread and will be consumed with bread
  Interventions: Dietary Supplement: Baobab spread

INTERVENTIONS:
Dietary Supplement: Baobab spread mixed with fermented brown seaweed — 5-day intake period
  Arms: Baobab spread mixed with fermented seaweed
Dietary Supplement: Baobab spread — 5-day intake period
  Arms: Baobab spread

SUMMARY:
The aim of this randomised, controlled, cross-over study is to investigate whether the intake of fermented brown seaweed can lower postprandial blood glucose levels and influence the composition of the gut microbiota in 25 healthy volunteers. Well-being and gastrointestinal symptoms as well as sensory properties of the products will also be evaluated using questionnaires.

At the screening visit, the subjects will be informed about the study procedures and inclusion/exclusion criteria will be checked. Informed consent will be signed by each subject before participating in the study. The participants will consume the active and control product, respectively, for 5 days with a 14-day wash-out period in between. Capillary blood samples will be drawn for glucose measurement at the first day of each 5-day intervention period. Faecal samples will be collected before and after each 5-day intervention period to analyse changes in gut microbial composition.

DETAILED DESCRIPTION:
Fermented seaweed is a sustainable food with increasing interest as an ingredient of a plant-based diet. Plant-based diets are gaining popularity both because of their health benefits and low-carbon footprint. Seaweed is a rich source of minerals, polyphenols and dietary fibres like xylans, carrageenan, fucoidan, laminarin and alginate. These bioactive compounds have been shown to exert positive effects on metabolic parameters, such as blood glucose and insulin, blood lipid profile and inflammatory markers and could therefore help in the prevention of cardiovascular diseases. Besides possible health benefits, fermentation of seaweed can offer potential advantages such as improved food safety and shelf life of non-dried seaweed as well as improved sensory properties.

The project aims to investigate the effects of fermented brown seaweed (Alaria Esculenta, also known as winged kelp) on glucose metabolism and its prebiotic potential in humans. A short-term pilot study (5-day intake period) will be conducted in young healthy subjects.

Twenty-five healthy subjects will be recruited to this study. This study will be a randomised controlled cross-over study where all participants will consume the test product and the control product for 5 days. In between each 5-day intervention period, there will be a wash-out period of 2 weeks.

At the first day of each 5-day intake period, the subjects have to come to the study centre in the morning in a fasting state. A test meal with the active product or control product containing each 50g of total carbohydrates will be served. Blood samples (finger-pricking) will be taken at fasting state (0 min) and at 15, 30, 45, 60, 90, 120, 150 and 180 min. The participants will then consume the product daily for 5 days at a dose of 2x 15g baobab with or without (control) 15% of the fermented seaweed. The product will be available as a spread in packages of 15g. After a wash-out period of 2 weeks, the participants will take the other product (cross-over design).

Faecal samples will be collected before and at the end of each 5-day intervention period. The questionnaire about well-being and gastrointestinal symptoms will be filled at home daily during each 5-day intervention. Also, a sensory questionnaire will be filled in at day 1 and 5 of intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age 20-40 years, at the time of signing the informed consent
* BMI 20-25 kg/m2
* Stable body weight (less than 5% difference during the last 3 months)
* Willing and able to give written informed consent for participating the study
* Willing to comply with all study procedures

Exclusion Criteria:

* Intake of antibiotics within 4 weeks prior to the start of the study
* Regular intake of probiotics and/or prebiotics within 4 weeks prior to the start of the study
* Tobacco use (smoking and/or snus)
* High alcohol intake: > 4 glasses daily
* Pregnancy or lactating
* Chronical disease (e.g., liver, kidney)
* Diabetes
* Gastrointestinal disease (ulcerative colitis, Crohn's disease, irritable bowel syndrome)
* Heart disease (within the last 12 months)
* Inflammatory disease (e.g. asthma, GI inflammatory diseases) and auto-immune disease
* Treatment with corticosteroids of significant degree
* Psychological disease of significant degree
* Cancer of significant difference
* Gastric-bypass operation
* Operation planned during the study period
* Known gluten intolerance and/or lactose intolerance
* Having allergies to the food components of the study, mustard and seafoods
* Known gluten intolerance, lactose intolerance, milk protein allergy or other food allergies
* Irregular diet (i.e., not eating 3 main meals daily) or special diet (e.g. vegan, low-carb high-fat, 5-2)
* Investigator considers the subject unlikely to comply with the study procedures, restrictions, and requirements

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood glucose | 0- 180 minutes (after intake of the study product)
  iAUC 0- 180 minutes

SECONDARY OUTCOMES:
Gut microbiota | Before and immediately after each 5-day intake period
  Total and Lactobacillus specific bacterial communities will be measured in fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Lieselotte Cloetens, Principal Investigator — Lund University
Locations (1):
- Aventure Clinical Trial Unit, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No